CLINICAL TRIAL: NCT04881656
Title: Evaluating the Impact of Telehealth-Based Autism Spectrum Disorder Assessments and Supports on Child and Caregiver Outcomes
Brief Title: Evaluating the Impact of Telehealth-Based ASD Assessments and Supports on Child and Caregiver Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1749700; UL1TR001860 (NIH)
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; telehealth
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIYH (Experimental): Help is in Your Hands is a series of online modules for parents with narrated videos of specific interactive strategies for supporting toddlers' communication development.
  Interventions: Other: Help is in Your Hands
- Comparison (No Intervention): No additional materials

INTERVENTIONS:
Other: Help is in Your Hands — HIIYH is a set of 16 online educational modules for caregivers of children with social-communication delays or elevated likelihood of ASD.
  Other Names: HIIYH
  Arms: HIIYH

SUMMARY:
The overall goal of this study is to evaluate telehealth and internet-based approaches to meet accessibility challenges for families with concerns about ASD in their infants. In this study, we will gather exploratory data related to the potential of two telehealth tools: 1) The Telehealth Evaluation of Development for Infants (TEDI); and 2) "Help is in Your Hands" (HIIYH), a set of video materials and information on interactive strategies parents can use to support their child's communication development. We will recruit families participating in an ongoing study using the TEDI (R21 HD100372, PI: Talbott) to evaluate infants' behavioral development. As families exit the parent TEDI study and enter the current study, we will ask parents to complete online questionnaires, and randomize them to either receive immediate access to additional online materials (HIIYH) for parents or no additional materials. After 12 weeks, parents will complete online questionnaires and all families will then be given access to the online materials. When children reach 30 months, we will collect additional questionnaires, complete a live telehealth behavioral session with toddlers and their caregivers, and conduct an exit interview with parents to gather feedback about their experience.

ELIGIBILITY:
Inclusion Criteria:

Previous enrollment in the parent R21 project (R21 HD100372, PI: Talbott).

Exclusion Criteria:

No previous enrollment in the parent R21 project (R21 HD100372, PI: Talbott).

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2033-05-31 (Estimated)

PRIMARY OUTCOMES:
Parent Stress Index 4th Edition, Short Form | Change from baseline at 12 weeks
  Mean Score
Parent Sense of Competence | Change from baseline at 12 weeks
  Mean Score
Telehealth Usability Questionnaire | Change from baseline at 12 weeks
  Mean Score

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Talbott, Ph.D., Principal Investigator — University of California Davis, MIND Institute
Locations (1):
- University of California Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/telehealth-evaluation-of-development-for-toddlers-372508/